CLINICAL TRIAL: NCT05445544
Title: A Multicenter Cohort Study on Maternal and Infant Microecology and New Targets for Pre-eclampsia Screening in China
Acronym: CALM2001
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Foshan Women's and Children's Hospital (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Hongwei Zhou, Proffessor, Zhujiang Hospital
Other Study IDs: CALM2001
Record Dates: First submitted 2022-06-20; First posted 2022-07-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Preeclampsia; Microbiome
Keywords: preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimen will include urines ,serums ,salivas, feces,vaginal swabs and placentas, cord bloods and amniotic fluids from the volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women and Follow-up of pregnant women's newborns: The pregnant woman is pregnant until she gives birth. The fecal ,serum,saliva,urine,vaginal secretions,umbilical cord blood,placenta and amniotic fluids who are were caesarean delivered will be collected
  Interventions: Other: Observational studies, The diagnosis was preeclampsia

INTERVENTIONS:
Other: Observational studies, The diagnosis was preeclampsia — Observational studies, The diagnosis was preeclampsia

SUMMARY:
major objective This multicenter, prospective cohort study aims at evaluating the predictive value of microbiome ,proteomics and serum markers in preeclampsia. secondary objective to evaluate the value of microbiome,proteomics and serum markers in assessing pregnancy outcome (complications during pregnancy and delivery, delivery) and neonatal prognosis.

DETAILED DESCRIPTION:
The volunteers will be recruited from the gestational women who come to the hospital before 14 weeks of gestation. After being informed about the potential risks, each volunteer giving written informed consent will be asked to complete a questionnaire. Then,urines ,serums and salivas as well as vaginal swabs and feces will be taken from each volunteer at gestational ages 11-14, 22-28, 32-34 weeks and delivery period .In delivery period,we will take placentas, cord bloods, amniotic fluids if it is possible. They will be followed up to two years after the child delivery (6 weeks,6 months,1 years and 2years after the child delivery) and do the same sampling who have preeclampsia during gestation. The salivas, vaginal swabs,placentas, amniotic fluids and feces will be to perform 16S rRNA(ribosomal ribonucleic acid) gene sequencing microecology assessment, Body fluid samples will be to perform peptidomics by MALDI-TOF(Matrix-Assisted Laser Desorption/ Ionization Time of Flight ) and metabonomics by mass spectrometer, combinations of mean arterial pressure (MAP), uterine artery pulsatile index , serum placental growth factor (PlGF) to estimate the patient-specific risk of pre-eclampsia (PE) .

ELIGIBILITY:
Inclusion Criteria:

* Aged >=18 years;
* Pregnancy woman;
* With a singleton pregnancy;
* Volunteer and receive regular antenatal examinations in the research centers;
* Volunteer to sign a written informed consent.

Exclusion Criteria:

* Concurrent with hypertension, diabetes, liver and kidney diseases, hematonosis and other serious diseases of pre-pregnancy women, including patients requiring long-term medication for primary diseases;
* With history of preeclampsia;
* Tumor patients concurrent with serious infection requiring long-term drug treatment;
* Pregnant women conceiving through in vitro fertilization;
* Multiple pregnancies;
* Patients with clear indications of medical pregnancy termination during early pregnancy;
* Any medical or non-medical conditions deemed inappropriate for study participation according to the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Preeclampsia is a condition in women during pregnancy
Study Population: All the patients in pregnancy will be eligible to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
microbiome | 34 months
  To evaluate the predictive value of microbiome in preeclampsia. To observe the changes of microbiome in pregnant women with preeclampsia from 11-14 weeks of gestation to two years postpartum.The microbial composition of the stool samples was determined by 16S rRNA (ribosomal ribonucleic acid) gene sequencing analysis and metagenomics.
proteomics | 34 months
  To evaluate the predictive value of proteomics in preeclampsia. To observe the changes of urine and serum proteomics in pregnant women with preeclampsia from 11-14 weeks of gestation to two years postpartum. proteomics is the large-scale study of small or big molecules, such as protein,polypeptide.
metabonomics | 34 months
  To evaluate the predictive value of metabonomics in preeclampsia. To observe the changes of serum metabonomics in pregnant women with preeclampsia from 11-14 weeks of gestation to two years postpartum. Metabolomics is the large-scale study of small molecules, such as fatty acids, bile acids, lipid mediators and others.

SECONDARY OUTCOMES:
microbiome | 10 months
  To evaluate the value of microbiome in assessing pregnancy outcome (complications during pregnancy and delivery, delivery) . To observe the changes of microbiome in pregnant women from 11-14 weeks of gestation to delivery.The microbial composition of the stool samples was determined by 16S rRNA (ribosomal ribonucleic acid) gene sequencing analysis and metagenomics.
proteomics | 10 months
  To evaluate the value of proteomics in assessing pregnancy outcome (complications during pregnancy and delivery, delivery) . To observe the changes of proteomics in pregnant women from 11-14 weeks of gestation to delivery.proteomics is the large-scale study of small or big molecules, such as protein,polypeptide.
metabonomics | 10 months
  To evaluate the value of metabonomics in assessing pregnancy outcome (complications during pregnancy and delivery, delivery) . To observe the changes of metabonomics in pregnant women from 11-14 weeks of gestation to delivery. Metabolomics is the large-scale study of small molecules, such as fatty acids, bile acids, lipid mediators and others.

CONTACTS AND LOCATIONS:
Overall Officials: hongwei zhou, Study Chair — Zhujiang Hospital
Locations (2):
- China (2):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Zhujiang hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen X, Li P, Liu M, Zheng H, He Y, Chen MX, Tang W, Yue X, Huang Y, Zhuang L, Wang Z, Zhong M, Ke G, Hu H, Feng Y, Chen Y, Yu Y, Zhou H, Huang L. Gut dysbiosis induces the development of pre-eclampsia through bacterial translocation. Gut. 2020 Mar;69(3):513-522. doi: 10.1136/gutjnl-2019-319101. Epub 2020 Jan 3. PMID 31900289